CLINICAL TRIAL: NCT06573255
Title: Assessment of Cardiopulmonary Fitness in Healthy Adults
Status: Recruiting | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Ebru Calik Kutukcu, Professor, Hacettepe University
Other Study IDs: GO 23/211
Record Dates: First submitted 2024-08-26; First posted 2024-08-27 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Healthy
Keywords: cardiorespiratory fitness

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Healthy group — Cardiopulmonary exercise test, respiratory function tests, respiratory muscle strength and physical activity assessment will be performed in this group.

SUMMARY:
This project was aimed to investigate cardiorespiratory fitness and the factors affecting cardiorespiratory fitness in healthy adults. The data obtained with this project will be normative values for the data obtained with CPET in healthy people.

DETAILED DESCRIPTION:
Cardiorespiratory fitness is one of the 'health-related physical fitness' components of physical fitness and can be expressed as 'the ability of the heart, lung and vascular system to deliver oxygen and nutrients to working muscles'. Cardiopulmonary exercise testing (CPET) is a common procedure used to assess cardiopulmonary fitness, identify physiological factors limiting exercise, identify potential therapeutic targets for these factors, and evaluate the effects of an intervention. Therefore, in this project, it was aimed to investigate cardiorespiratory fitness and the factors affecting cardiorespiratory fitness in healthy adults. The data obtained with this project will be normative values for the data obtained with CPET in healthy people.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years of age,
* Volunteering to participate in the study,
* Co-operation,
* Being able to ambulate.

Exclusion Criteria:

* Having any known respiratory, cardiac, neurological or other internal disease or malignant disease,
* Having any problem or musculoskeletal system disorder that prevents walking,
* To have undergone any surgery within the last six months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will include healthy adult subjects without any known internal disease.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-04-18 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Cardiorespiratory Fitness | This test takes 15 to 20 minutes.
  In this parameter, which is assessed by cardiopulmonary exercise testing, the oxygen consumption measured during the test and the workload achieved in the test will be taken into consideration.

SECONDARY OUTCOMES:
Respiratory Function Test | This test takes 3 to 5 minutes.
  The pulmonary function test is a test that assesses respiratory function by performing certain manoeuvres.
Respiratory Muscle Strength Test | This test takes 3 to 5 minutes.
  Inspiratory and expiratory muscle strengths will be measured separately by breathing manoeuvres.
Physical Activity | This questionnaire takes 1 minute.
  Physical activity level will be measured with International Physical Activity Questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Ebru Calik Kutukcu, PhD, Principal Investigator — Hacettepe Univesity
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided